CLINICAL TRIAL: NCT05113732
Title: Association of Cognition With Functional Mobility in People With Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kübra Nur Menengiç, Student of PhD, Istanbul University - Cerrahpasa
Other Study IDs: IUC-PT
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Alzheimer Dementia; Alzheimer's Disease; Dementia, Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to investigate relationship between cognitive function and functional mobility in Alzheimer's disease.

DETAILED DESCRIPTION:
Our hypothesis is that the decrease in cognitive function in individuals with Alzheimer's disease is associated with the level of functional mobility. Sociodemographic information of participants will be recorded. Cognition will assessed with Montreal Cognitive Assessment (MoCA), global score and MoCA's visuospatial executive functions, naming, attention, language, abstract thinking, delayed recall, orientation sub-scores will recorded. Functional mobility will assessed Timed Up and Go Test and 5 Times Sit&Stand Test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Alzheimer's disease according to the National Institute of --Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease (NINCDS-ADRDA) criteria,
* Over 65 years old,
* Cases who could understand the instructions given in Turkish were included in the study,
* Having ambulation skill independently or with walking aid.

Exclusion Criteria:

* Dementia with Lewy bodies, frontotemporal dementia and one of the other types of dementia,
* Having a pulmonary, neurological, musculoskeletal or rheumatological disease that may prevent exercise,
* Unstable medical condition (uncontrolled diabetes or hypertension, deep vein thrombosis, etc.),
* Subjects with visual or auditory deficits or behavioral problems that would make communication difficult were not included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with Alzheimer's disease
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assesment (MoCA) | Baseline
  MoCA assesses cognitive skills such as visuospatial / executive functioning, object naming, memory, attention, language, abstraction, orientation. Higher scores reflect the better performance.
Timed Up and Go Test | Baseline
  Timed Up and Go Test measures the level of functional mobility skills and, assess fall risk and balance. The time elapsed between standing up from the sitting position, walking the distance of 3 meters, coming back and sitting back on the chair is recorded. The shorter time reflect the better performance.
5 Time Sit to Stand Test | Baseline
  5 Time Sit to Stand Test measures the level of functional mobility skills and, assess fall risk and lower extremity strength. The test measures the time taken to stand five times from a sitting position as quickly as possible. The shorter time reflect the better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)